CLINICAL TRIAL: NCT05958888
Title: Visual Attention to Text and Pictorial Food Labels: An Eye Tracking Experiment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 23-0659; K01HL147713 (NIH)
Record Dates: First submitted 2023-07-12; First posted 2023-07-25 (Actual); Results first posted 2024-08-13 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2023-10

CONDITIONS: Health Behavior
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Intervention Model Description: All participants will see the same 4 labels (3 sodium labels [text only, text + icon, and text + pictorial] and a control bar code label) in a random order.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Front of package food label (Experimental): 4 labels (3 sodium labels, 1 control barcode label) are shown on an image of a soup can
  Interventions: Behavioral: Text only sodium label; Behavioral: Icon sodium label; Behavioral: Pictorial sodium label; Behavioral: Barcode label

INTERVENTIONS:
Behavioral: Text only sodium label — "Warning: High in sodium." is shown in a black square label on the can of soup.
Behavioral: Icon sodium label — "Warning: High in sodium." is shown beneath a yellow triangle icon with an exclamation mark all in a black square label on the can of soup.
Behavioral: Pictorial sodium label — "Warning: High in sodium." is shown beneath an image of a spilled salt shaker, all in a black square label on the can of soup.
Behavioral: Barcode label — Barcode is shown in white square label on the can of soup

SUMMARY:
The goal of this study is to examine attention elicited by icon, text-only, and control front-of-package food labels. The study also aims to explore whether English language proficiency moderates the impact of icon vs. text-only labels on attention.

DETAILED DESCRIPTION:
In this study, participants will attend one in-person visit, lasting approximately 15 minutes after signing informed consent. First participants will complete an eye tracking task where their attention to study stimuli is measured objectively via an eye tracker (i.e., eye tracking task). The eye tracking task will take ~5 minutes. Then, participants will complete a brief ~10 minute self-administered survey on a computer.

ELIGIBILITY:
Inclusion Criteria:

* Adult aged 18 or older
* Self-identifies as Hispanic or Latino

Exclusion Criteria:

* Less than 18 years old
* Does not identify as Hispanic or Latino
* Has one of the following conditions: (Wears bifocals, glaucoma, permanently dilated pupils, eye implants [artificial lenses, not contact lenses], less than 2 eyes, or blindness)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2023-08-02 (Actual); Primary Completion 2023-09-29 (Actual); Study Completion 2023-09-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marissa Hall, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with the University of North Carolina (UNC).
Supporting Information: SAP, Analytic Code
Time Frame: Data will be available 9 months after and up to 10 years following publication.
Access Criteria: The investigator has approved IRB, IEC, or REB and an executed data use/sharing agreement with UNC.

RESULTS

PARTICIPANT FLOW:
Groups:
- Front of Package Food Label: Participants view 4 labels (3 sodium labels, 1 control barcode label) on a soup can image in a random order with a washout in between each label viewing. The washout includes instructions to click forward at participants' own pace to view the next label.
  Text only sodium label: "Warning: High in sodium." is shown in a black square label on the can of soup.
  Icon sodium label: "Warning: High in sodium." is shown beneath a yellow triangle icon with an exclamation mark all in a black square label on the can of soup.
  Pictorial sodium label: "Warning: High in sodium." is shown beneath an image of a spilled salt shaker, all in a black square label on the can of soup.
  Barcode label: Barcode is shown in white square label on the can of soup
Period: First Label Viewing (Self-paced)
Arm/Group | Front of Package Food Label
Started | 63
Text Only Sodium Label | 17
Icon Sodium Label | 18
Pictorial Sodium Label | 11
Barcode Label | 17
Completed | 63
Not Completed | 0
Period: Washout (Self-paced)
Arm/Group | Front of Package Food Label
Started | 63
Text Only Sodium Label | 17
Icon Sodium Label | 18
Pictorial Sodium Label | 11
Barcode Label | 17
Completed | 63
Not Completed | 0
Period: Second Label Viewing (Self-paced)
Arm/Group | Front of Package Food Label
Started | 63
Text Only Sodium Label | 15
Icon Sodium Label | 13
Pictorial Sodium Label | 22
Barcode Label | 13
Completed | 63
Not Completed | 0
Period: Washout (Self Paced)
Arm/Group | Front of Package Food Label
Started | 63
Text Only Sodium Label | 15
Icon Sodium Label | 13
Pictorial Sodium Label | 22
Barcode Label | 13
Completed | 63
Not Completed | 0
Period: Third Label Viewing (Self-paced)
Arm/Group | Front of Package Food Label
Started | 63
Text Only Sodium Label | 21
Icon Sodium Label | 10
Pictorial Sodium Label | 14
Barcode Label | 18
Completed | 63
Not Completed | 0
Period: Washout (Self Paced)
Arm/Group | Front of Package Food Label
Started | 63
Text Only Sodium Label | 21
Icon Sodium Label | 10
Pictorial Sodium Label | 14
Barcode Label | 18
Completed | 63
Not Completed | 0
Period: Fourth Label Viewing (Self-paced)
Arm/Group | Front of Package Food Label
Started | 63
Text Only Sodium Label | 10
Icon Sodium Label | 22
Pictorial Sodium Label | 16
Barcode Label | 15
Completed | 63
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Front of Package Food Label
Number analyzed (Participants) | 63
Age, Continuous [Mean (Standard Deviation); unit: years] | 34 (10)
Age, Customized [Count of Participants; unit: Participants]
  Age categories: 18-25 years | 11
  Age categories: 26-34 years | 22
  Age categories: 35-44 years | 20
  Age categories: 45-54 years | 8
  Age categories: Over 55 years | 2
Sex/Gender, Customized [Count of Participants; unit: Participants] — Population: Reporting of gender was optional and 1 participant did not provide.
  Participants
    Gender identity: number analyzed (Participants) | 62
    Gender identity: Woman | 47
    Gender identity: Man | 15
    Gender identity: Non-binary | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Mexican, Mexican American, Chicano | 24
  Ethnicity: Puerto Rican | 5
  Ethnicity: Cuban | 0
  Ethnicity: Another Hispanic, Latino, or Spanish origin | 34
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 63

OUTCOME MEASURES:

1. Primary Outcome: Amount of Time Spent Looking at the Front-of-package Sodium Label (i.e., Dwell Time)
Description: This outcome will be measured using eye tracking technology.
Time Frame: During ~5-minute eye tracking task, as part of a one-time study visit lasting ~30 minutes
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Front of Package Food Label
Number analyzed (Participants) | 63
seconds
  Barcode Control | .96 (.88)
  Text | 1.94 (1.23)
  Icon | 2.34 (2.43)
  Graphic | 2.58 (1.53)
Statistical Analysis 1: Comparison: Front of Package Food Label; Text vs. Control; Test type: Superiority; p < 0.001, Mixed Models Analysis — p-values were adjusted for multiple comparisons using the Bonferroni-Holm method, correcting for six tests within each outcome. The a priori threshold for statistical significance was p<0.05; Mean Difference (Final Values) = .99, Standard Error of Mean .20
Statistical Analysis 2: Comparison: Front of Package Food Label; Icon vs. Control; Test type: Superiority; p < 0.001, Mixed Models Analysis — p-values were adjusted for multiple comparisons using the Bonferroni-Holm method, correcting for six tests within each outcome.The a priori threshold for statistical significance was p<0.05; Mean Difference (Final Values) = 1.39, Standard Error of Mean .20
Statistical Analysis 3: Comparison: Front of Package Food Label; Graphic vs. Control; Test type: Superiority; p < .001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 1.62, Standard Error of Mean .20
Statistical Analysis 4: Comparison: Front of Package Food Label; Icon vs. Text; Test type: Superiority; p = .10, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = .40, Standard Error of Mean .20
Statistical Analysis 5: Comparison: Front of Package Food Label; Graphic vs. Text; Test type: Superiority; p = .01, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = .63, Standard Error of Mean .20
Statistical Analysis 6: Comparison: Front of Package Food Label; Graphic vs. Icon; Test type: Superiority; p = .25, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = .23, Standard Error of Mean .20

2. Secondary Outcome: Number of Times Looking at the Front-of-package Sodium Label (i.e., Fixation Count)
Description: This outcome will be measured using eye tracking technology.
Time Frame: During ~5-minute eye tracking task, as part of a one-time study visit lasting ~30 minutes
Measure: Mean (Standard Deviation); unit: fixation
Arm/Group | Front of Package Food Label
Number analyzed (Participants) | 63
fixation
  Barcode Control | 5 (4)
  Text | 9 (5)
  Icon | 11 (8)
  Graphic | 13 (6)
Statistical Analysis 1: Comparison: Front of Package Food Label; Text vs. Control; Test type: Superiority; p < .001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 4, Standard Error of Mean .85
Statistical Analysis 2: Comparison: Front of Package Food Label; Icon vs. Control; Test type: Superiority; p < .001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 6, Standard Error of Mean .85
Statistical Analysis 3: Comparison: Front of Package Food Label; Graphic vs. Control; Test type: Superiority; p < .001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 8, Standard Error of Mean .85
Statistical Analysis 4: Comparison: Front of Package Food Label; Icon vs. Text; Test type: Superiority; p = .12, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 1, Standard Error of Mean .85
Statistical Analysis 5: Comparison: Front of Package Food Label; Graphic vs. Text; Test type: Superiority; p < .001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 3, Standard Error of Mean .85
Statistical Analysis 6: Comparison: Front of Package Food Label; Graphic vs. Icon; Test type: Superiority; p = .04, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 2, Standard Error of Mean .85

3. Secondary Outcome: Time to First Fixation on the Front-of-package Sodium Label
Description: This outcome will be measured using eye tracking technology.
Time Frame: During ~5-minute eye tracking task, as part of a one-time study visit lasting ~30 minutes
Population: There were missing data for 1 participant.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Front of Package Food Label
Number analyzed (Participants) | 62
seconds
  Barcode Control | .87 (1.60)
  Text | .31 (.45)
  Icon | .52 (1.30)
  Graphic | .27 (.36)
Statistical Analysis 1: Comparison: Front of Package Food Label; Text vs. Control; Test type: Superiority; p = .01, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -.56, Standard Error of Mean .19
Statistical Analysis 2: Comparison: Front of Package Food Label; Icon vs. Control; Test type: Superiority; p = .23, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -.35, Standard Error of Mean .19
Statistical Analysis 3: Comparison: Front of Package Food Label; Graphic vs. Control; Test type: Superiority; p = .01, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -.59, Standard Error of Mean .19
Statistical Analysis 4: Comparison: Front of Package Food Label; Icon vs. Text; Test type: Superiority; p = .58, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = .21, Standard Error of Mean .19
Statistical Analysis 5: Comparison: Front of Package Food Label; Graphic vs. Text; Test type: Superiority; p = .85, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -.03, Standard Error of Mean .19
Statistical Analysis 6: Comparison: Front of Package Food Label; Graphic vs. Icon; Test type: Superiority; p = .58, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -.24, Standard Error of Mean .19

4. Secondary Outcome: Dwell Time on "Natural" Claim
Description: This outcome will be measured using eye tracking technology.
Time Frame: During ~5-minute eye tracking task, as part of a one-time study visit lasting ~30 minutes
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Front of Package Food Label
Number analyzed (Participants) | 63
seconds
  Barcode Control | .90 (.96)
  Text | .91 (1.00)
  Icon | .87 (.87)
  Graphic | .74 (.78)
Statistical Analysis 1: Comparison: Front of Package Food Label; Text vs. Control; Test type: Superiority; p > .99, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = .01, Standard Error of Mean .10
Statistical Analysis 2: Comparison: Front of Package Food Label; Icon vs. Control; Test type: Superiority; p > .99, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -.03, Standard Error of Mean .10
Statistical Analysis 3: Comparison: Front of Package Food Label; Graphic vs. Control; Test type: Superiority; p = .47, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -.16, Standard Error of Mean .10
Statistical Analysis 4: Comparison: Front of Package Food Label; Icon vs. Text; Test type: Superiority; p > .99, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -.04, Standard Error of Mean .10
Statistical Analysis 5: Comparison: Front of Package Food Label; Graphic vs. Text; Test type: Superiority; p = .45, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -.17, Standard Error of Mean .10
Statistical Analysis 6: Comparison: Front of Package Food Label; Graphic vs. Icon; Test type: Superiority; p = .70, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -.13, Standard Error of Mean .10

5. Secondary Outcome: Self-reported Attention to the Front-of-package Sodium Label
Description: Assessed with 1 item for each label type. Response options will range from 1 to 5. Higher scores indicate more attention.
Time Frame: During ~10 minute online survey, as part of one-time study visit lasting ~30 minutes
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Front of Package Food Label
Number analyzed (Participants) | 63
score on a scale
  Barcode Control | 2.40 (1.20)
  Text | 3.29 (.96)
  Icon | 4.16 (1.02)
  Graphic | 4.10 (.93)
Statistical Analysis 1: Comparison: Front of Package Food Label; Text vs. Control; Test type: Superiority; p < .001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = .89, Standard Error of Mean .17
Statistical Analysis 2: Comparison: Front of Package Food Label; Icon vs. Control; Test type: Superiority; p < .001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 1.76, Standard Error of Mean .17
Statistical Analysis 3: Comparison: Front of Package Food Label; Graphic vs. Control; Test type: Superiority; p < .001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 1.70, Standard Error of Mean .17
Statistical Analysis 4: Comparison: Front of Package Food Label; Icon vs. Text; Test type: Superiority; p < .001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = .87, Standard Error of Mean .17
Statistical Analysis 5: Comparison: Front of Package Food Label; Graphic vs. Text; Test type: Superiority; p < .001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = .81, Standard Error of Mean .17
Statistical Analysis 6: Comparison: Front of Package Food Label; Graphic vs. Icon; Test type: Superiority; p = .72, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -.06, Standard Error of Mean .17

6. Secondary Outcome: Perceived Message Effectiveness of the Front-of-package Sodium Label
Description: Assessed with 3 items for each label type. Response options will range from 1 to 5. Higher scores indicate greater perceived message effectiveness.
Time Frame: During ~10 minute online survey, as part of one-time study visit lasting ~30 minutes
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Front of Package Food Label
Number analyzed (Participants) | 63
score on a scale
  Barcode Control | 1.74 (.98)
  Text | 3.47 (1.01)
  Icon | 4.13 (.91)
  Graphic | 3.85 (.94)
Statistical Analysis 1: Comparison: Front of Package Food Label; Text vs. Control; Test type: Superiority; p < .001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 1.73, Standard Error of Mean .14
Statistical Analysis 2: Comparison: Front of Package Food Label; Icon vs. Control; Test type: Superiority; p < .001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 2.39, Standard Error of Mean .14
Statistical Analysis 3: Comparison: Front of Package Food Label; Graphic vs. Control; Test type: Superiority; p < .001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 2.11, Standard Error of Mean .14
Statistical Analysis 4: Comparison: Front of Package Food Label; Icon vs. Text; Test type: Superiority; p < .001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = .66, Standard Error of Mean .14
Statistical Analysis 5: Comparison: Front of Package Food Label; Graphic vs. Text; Test type: Superiority; p = .01, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = .38, Standard Error of Mean .14
Statistical Analysis 6: Comparison: Front of Package Food Label; Graphic vs. Icon; Test type: Superiority; p = .04, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -.28, Standard Error of Mean .14

7. Secondary Outcome: Understandability of Front-of-package Sodium Label
Description: 1 item for each label type. Response options will range from 1 to 5. Higher scores indicate more understandability.
Time Frame: During ~10 minute online survey, as part of one-time study visit lasting ~30 minutes
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Front of Package Food Label
Number analyzed (Participants) | 63
score on a scale
  Barcode Control | 3.41 (1.23)
  Text | 4.00 (.93)
  Icon | 4.22 (.87)
  Graphic | 4.13 (.98)
Statistical Analysis 1: Comparison: Front of Package Food Label; Text vs. Control; Test type: Superiority; p < .001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = .59, Standard Error of Mean .15
Statistical Analysis 2: Comparison: Front of Package Food Label; Icon vs. Control; Test type: Superiority; p < .001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = .81, Standard Error of Mean .15
Statistical Analysis 3: Comparison: Front of Package Food Label; Graphic vs. Control; Test type: Superiority; p < .001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = .71, Standard Error of Mean .15
Statistical Analysis 4: Comparison: Front of Package Food Label; Icon vs. Text; Test type: Superiority; p = .43, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = .22, Standard Error of Mean .15
Statistical Analysis 5: Comparison: Front of Package Food Label; Graphic vs. Text; Test type: Superiority; p = .81, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = .13, Standard Error of Mean .15
Statistical Analysis 6: Comparison: Front of Package Food Label; Graphic vs. Icon; Test type: Superiority; p = .81, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -.10, Standard Error of Mean .15

ADVERSE EVENTS:
Time Frame: From the time of signing informed consent, through study completion, a total of up to 30 minutes.
Groups:
- Text Only Sodium Label: Participants are shown on an image of a soup can bearing a text only sodium label: "Warning: High in sodium." is shown in a black square label on the can of soup.
- Icon Sodium Label: Participants are shown on an image of a soup can bearing an icon sodium label: "Warning: High in sodium." is shown beneath a yellow triangle icon with an exclamation mark all in a black square label on the can of soup.
- Pictorial Sodium Label: Participants are shown on an image of a soup can bearing a pictorial sodium label: "Warning: High in sodium." is shown beneath an image of a spilled salt shaker, all in a black square label on the can of soup.
- Barcode Label: Participants are shown on an image of a soup can bearing a barcode label: Barcode is shown in white square label on the can of soup
Arm/Group | Text Only Sodium Label | Icon Sodium Label | Pictorial Sodium Label | Barcode Label
All-Cause Mortality (participants affected / at risk) | 0/63 | 0/63 | 0/63 | 0/63
Serious Adverse Events (participants affected / at risk) | 0/63 | 0/63 | 0/63 | 0/63
Other Adverse Events (participants affected / at risk) | 0/63 | 0/63 | 0/63 | 0/63

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-06-24): https://cdn.clinicaltrials.gov/large-docs/88/NCT05958888/Prot_SAP_001.pdf
  • Informed Consent Form (2023-05-23): https://cdn.clinicaltrials.gov/large-docs/88/NCT05958888/ICF_000.pdf